CLINICAL TRIAL: NCT01029717
Title: A Randomised Controlled Trial Comparing the Effectiveness of Heparin Bonded or Antibiotic Impregnated Central Venous Catheters (CVCs) With Standard CVCs for the Prevention of Hospital Acquired Blood Stream Infection in Children
Brief Title: CATCH - Catheter Infections in Children
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Institute of Child Health (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 08EB20
Record Dates: First submitted 2009-12-09; First posted 2009-12-10 (Estimated); Last update posted 2022-03-03 (Actual); Status verified 2022-02

CONDITIONS: Catheter-related Infections
Keywords: Central Venous Catheters; blood stream infection; children, intensive care; Heparin bonded; antibiotic coated; Children in Paediatric Intensive Care Unit
MeSH Terms: conditions — Catheter-Related Infections

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- Standard polyurethane Central Venous Catheter (Experimental): Standard polyurethane Central Venous Catheter
  All CVCs used in the trial are CE marked medical devices used for their intended purpose.
  Interventions: Device: Standard polyurethane Central Venous Catheter
- Antibiotic impregnated polyurethane CVC (Active Comparator): Antibiotic impregnated polyurethane CVC (minocycline and rifampicin)
  All CVCs used in the trial are CE marked medical devices used for their intended purpose.
  Interventions: Device: Antibiotic impregnated polyurethane CVC (minocycline and rifampicin)
- Heparin bonded polyurethane CVC (Active Comparator): Heparin bonded polyurethane CVC
  All CVCs used in the trial are CE marked medical devices used for their intended purpose.
  Interventions: Device: Heparin bonded polyurethane CVC

INTERVENTIONS:
Device: Standard polyurethane Central Venous Catheter — Standard polyurethane Central Venous Catheter, All CVCs used in the trial are CE marked medical devices used for their intended purpose.
  Arms: Standard polyurethane Central Venous Catheter
Device: Antibiotic impregnated polyurethane CVC (minocycline and rifampicin) — Antibiotic impregnated polyurethane CVC (minocycline and rifampicin. All CVCs used in the trial are CE marked medical devices used for their intended purpose.
  Arms: Antibiotic impregnated polyurethane CVC
Device: Heparin bonded polyurethane CVC — Heparin bonded polyurethane CVC. All CVCs used in the trial are CE marked medical devices used for their intended purpose.
  Arms: Heparin bonded polyurethane CVC

SUMMARY:
Most children admitted to paediatric intensive care units (PICU) need to have medicines given to them into their veins using a narrow tube, so they do not need repeated injections. This tube is called a central venous catheter. Occasionally these catheters can cause infections in the blood and sometimes the tubes can get blocked by small blood clots.

Some intensive care units already use antibiotic or heparin coated catheters, but there is no proof that these are better than the standard ones at preventing infections. Most of the PICU's in this country use standard lines. The only way to find out for certain is to compare children who are given antibiotic or heparin coated catheters with those who are given standard ones in a clinical trial. Because we do not know which type of catheter is best, the type of catheter each child receives in the study will be decided randomly by chance.

Each child in the trial will have the same chance of getting any of these three catheters:

* Standard central venous catheter (not coated).
* Heparin coated central venous catheter. Heparin is a medicine that can stop blood from clotting and might stop the tubes being blocked and infections in the blood.
* Antibiotic coated central venous catheter. Antibiotics can be used to kill bacteria which cause the infections.

The aim of this study is to see how the three types of catheters compare in reducing the amount of blood infections in children. We will also look at the costs involved. We hope to recruit 1200 children in the UK over 2 years. We hope that the information we get from this study will guide policy about purchasing impregnated Central Venous Catheters across the NHS and thereby improve treatment for children in the future.

ELIGIBILITY:
Inclusion Criteria:

* Weighing ≥3kg and less than 16 years of age;
* Admitted to or being prepared for admission to an intensive care unit participating in the trial;
* Require insertion of a polyurethane CVC as part of good clinical management;
* Require one of the CVC sizes available to the trial (see Appendix A for the list of CVCs);
* Expected to require a CVC for at least 3 days;
* Appropriate consent obtained (prospective consent for elective surgical patients, deferred consent for emergency admission patients).

Max Age: 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 1859 (Actual)
Dates: Start 2010-12 (Actual); Primary Completion 2012-11 (Actual); Study Completion 2012-11 (Actual)

PRIMARY OUTCOMES:
The primary outcome will be time to first blood stream infection defined by a positive blood culture from a sample that was clinically indicated and taken more than 48 hours after CVC insertion and up to 48 hours after CVC removal. | 48 HOURS

CONTACTS AND LOCATIONS:
Overall Officials: Ruth Gilbert, Professor, Study Director — Institute of Child Health
Locations (1):
- Institute of Child Health, London, United Kingdom

REFERENCES:
- [Background] Pierce CM, Wade A, Mok Q. Heparin-bonded central venous lines reduce thrombotic and infective complications in critically ill children. Intensive Care Med. 2000 Jul;26(7):967-72. doi: 10.1007/s001340051289. PMID 10990114
- [Result] Harron K, Mok Q, Dwan K, Ridyard CH, Moitt T, Millar M, Ramnarayan P, Tibby SM, Muller-Pebody B, Hughes DA, Gamble C, Gilbert RE. CATheter Infections in CHildren (CATCH): a randomised controlled trial and economic evaluation comparing impregnated and standard central venous catheters in children. Health Technol Assess. 2016 Mar;20(18):vii-xxviii, 1-219. doi: 10.3310/hta20180. PMID 26935961
- [Derived] Harron K, Woolfall K, Dwan K, Gamble C, Mok Q, Ramnarayan P, Gilbert R. Deferred Consent for Randomized Controlled Trials in Emergency Care Settings. Pediatrics. 2015 Nov;136(5):e1316-22. doi: 10.1542/peds.2015-0512. Epub 2015 Oct 5. PMID 26438711